CLINICAL TRIAL: NCT00230516
Title: A Randomized, Open-Label, Comparative, Two-Treatment, Crossover Study of 24-hour Intragastric pH Profiles of Esomeprazole 40 mg and Lansoprazole 30 mg in Healthy Volunteer Subjects on Days 1 and 5 of Intravenous Treatment
Brief Title: Study of 24-hour Intragastric pH Profiles of Esomeprazole 40 mg and Lansoprazole 30 mg in Healthy Volunteer Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D9612L00080
Record Dates: First submitted 2005-09-28; First posted 2005-10-03 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: N/A this study is being conducted with healthy volunteers
MeSH Terms: interventions — Esomeprazole; Lansoprazole

INTERVENTIONS:
Drug: Nexium
Drug: Prevacid

SUMMARY:
This study is intended to evaluate whether intravenous (iv) esomeprazole (Nexium® ) offers better intragastric acid suppression than iv lansoprazole (Prevacid ®

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-70 years of age
* Participants can be male or female
* Women that are able to have children must have a negative pregnancy test.

Exclusion Criteria:

* Involvement in or planning of this study
* Participation in another clinical study within 28 days of this one
* For women, pregnancy or attempting to become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare the pharmacodynamic efficacy in controlling intragastric pH of esomeprazole 40mg and lansoprazole 30mg on Day 5 of once daily IV administration to healthy volunteers.

SECONDARY OUTCOMES:
Secondary Outcomes will compare additional efficacy and safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, Los Angeles, California
  - Research Site, Oklahoma City, Oklahoma